CLINICAL TRIAL: NCT03738514
Title: Comparison Of Efficacy Of Dentifrice Containing 5% Fluorocalcium Phosphosilicate With Dentifrice Containing Potassium Nitrate And Placebo On Dentinal Hypersensitivity: A Triple Masked Randomized Controlled Clinical Trial
Brief Title: Comparison of Efficacy of 5% Fluorocalcium Phosphosilicate Dentifrice and Potassium Nitrate Dentifrice on Dentinal Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Collaborators: Group Pharma (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Head and Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/Ph.D/5/2016-2017
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Dentinal Hypersensitivity
Keywords: Dentinal Hypersensitivity; Visual Analogue Score

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): dentifrice containing 5% fluorocalcium phospho silicate prescribed and VAS score assessed at Baseline, 2 weeks, 6 weeks.
  Interventions: Other: 5% fluorocalcium phosphosilicate dentifrice
- Group 2 (Sham Comparator): dentifrice containing 5% potassium nitrate prescribed and VAS score assessed at Baseline, 2weeks, 6 weeks .
  Interventions: Other: 5% potassium nitrate dentifrice
- Group 3 (Placebo Comparator): dentifrice without the active ingredient prescribed and VAS score assessed at Baseline, 2weeks, 6 weeks .
  Interventions: Other: Placebo dentrifice

INTERVENTIONS:
Other: 5% fluorocalcium phosphosilicate dentifrice — dentifrice containing 5% fluorocalcium phosphosilicate and VAS score assessed at Baseline, 2 weeks, 6 weeks
  Arms: Group 1
Other: 5% potassium nitrate dentifrice — 5% potassium nitrate dentifrice and VAS score assessed at Baseline, 2weeks, 6 weeks.
  Arms: Group 2
Other: Placebo dentrifice — placebo dentifrice and VAS score assessed at Baseline, 2weeks, 6 weeks
  Arms: Group 3

SUMMARY:
Aim of this study was to assess and compare the efficacy of a dentifrice containing 5% fluoro calcium phosphosilicate and dentifrice containing potassium nitrate on Dentinal Hypersensitivity (DH) compared to a placebo over a period of 6 weeks.

DETAILED DESCRIPTION:
A total of 120 subjects were divided into 3 groups randomly. Group 1 was given the dentifrice containing 5% fluoro calcium phosphosilicate ,Group 2 was given the dentifrice containing potassium nitrate and group 3 was given placebo. Sensitivity scores (VAS score) were recorded at baseline, 2 weeks, 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The volunteers selected at baseline were in good general health and should have at least 20 natural permanent teeth and history of hypersensitivity to hot, cold, sour stimuli on at least two teeth with a VAS score of ≥4.

Exclusion Criteria:

* Patients with active cervical caries or deep abrasion requiring cervical filling, chipped teeth or fractured cusps, tender tooth in same quadrant as the hypersensitive teeth, Subjects using any type of desensitizing paste or desensitizing therapy for last 6 months, Pregnant/ lactating women or subjects with history of chronic use of anti-inflammatory and analgesic medications were excluded.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale score for Dentinal Hypersensitivity | Change in VAS score from Baseline to 12 weeks
  Based on a 10-cm VAS score which was used to measure tooth sensitivity, a pain-free response was allotted a score of zero whereas a score of 10 was given to subjects with excruciating pain or discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Avani R Pradeep, MDS, Principal Investigator — GDCRI, Bangalore, INDIA
Locations (1):
- Department of Periodontics, GDCRI Bangalore, Bangalore, Karnataka, India